CLINICAL TRIAL: NCT00003358
Title: Phase I Trial Intraperitoneal Cisplatin With Intraperitoneal Gemcitabine in Patients With Epithelial Ovarian Carcinoma
Brief Title: Cisplatin and Gemcitabine in Treating Patients With Refractory or Recurrent Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-129; MSKCC-97129; NCI-H98-0016
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Drug Therapy; Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: chemotherapy
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of cisplatin plus gemcitabine in treating patients with refractory or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of intraperitoneal (IP) gemcitabine given in combination with IP cisplatin in patients with refractory or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer. II. Determine the safety of this regimen in this patient population. III. Determine the pharmacokinetics of IP gemcitabine administered with IP cisplatin.

OUTLINE: This is a dose escalation study of gemcitabine. Patients receive intraperitoneal cisplatin on day 1 plus intraperitoneal gemcitabine on days 1, 8, and 15. No treatment will be given on day 22. Courses are repeated every 4 weeks. Patients receive up to 4 courses of therapy. Dose escalation of gemcitabine continues in cohorts of 3 patients until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 6 patients experience dose limiting toxicity (DLT). Patients are followed every 3 months for 2 years, then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 3-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically documented epithelial ovarian carcinoma or fallopian tube cancer or primary peritoneal cancer following initial cytoreductive surgery and chemotherapy with at least one cisplatin based chemotherapy regimen Must have undergone a second assessment procedure (laparoscopy or laparotomy) within 8 weeks of protocol entry, and have confirmation of residual disease no greater than 1.0 cm at the end of the procedure

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 3 times upper limit of normal (ULN) SGOT less than 3 times ULN Alkaline phosphatase less than 3 times ULN Renal: Creatinine less than 1.6 mg/dL Creatinine clearance at least 50 mL/min Other: Must have a functioning implanted subcutaneous intraperitoneal catheter No neuropathy of grade III or greater from prior chemotherapy No contraindication to intraperitoneal therapy e.g., intraabdominal infection or widespread adhesions

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1998-01; Primary Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Sabbatini P, Aghajanian C, Leitao M, Venkatraman E, Anderson S, Dupont J, Dizon D, O'Flaherty C, Bloss J, Chi D, Spriggs D. Intraperitoneal cisplatin with intraperitoneal gemcitabine in patients with epithelial ovarian cancer: results of a phase I/II Trial. Clin Cancer Res. 2004 May 1;10(9):2962-7. doi: 10.1158/1078-0432.ccr-03-0486. PMID 15131031